CLINICAL TRIAL: NCT02644083
Title: Modulation of Cerebral Grey Matter High Energy Phosphate Metabolites in Multiple Sclerosis by Dimethyl Fumarate
Brief Title: Tecfidera and MRI for Brain Energy in MS
Status: Terminated | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Rebecca Spain, Dr Rebecca Spain, MD, MSPH, Oregon Health and Science University
Other Study IDs: IRB 11364
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dimethyl fumarate
  Other Names: Tecfidera

SUMMARY:
The primary objective of this study is to test the hypothesis that DMF can improve mitochondrial function in the brain of people with MS. The investigators will assess mitochondrial function in the cerebral grey matter by measuring PCr and ATP by 31P magnetic resonance spectroscopy (MRS) and NAA in NAWM by 1H MRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS by 2010 McDonald criteria
* Relapsing clinical course
* Ages 18-55
* Laboratory values that allow initiation of dimethyl fumarate (Tecfidera)

Exclusion Criteria:

* Systemic disease associated with cerebrovascular disease (e.g. diabetes mellitus, hypertension, hyperlipidemia, coronary heart disease)
* Treatment with corticosteroids or disease-modifying therapies (interferon beta, glatiramer acetate, natalizumab, fingolimod, teriflunomide) within 30 days of the first baseline MRI scan.
* Treatment at any time with mitoxantrone, cyclophosphamide, or any other long acting immunosuppressant
* Prior treatment of greater than 1 month at any time with DMF
* Inability to tolerate MRI procedures
* Pregnant/breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 21 patients with a diagnosis of relapsing-remitting multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Changes in phosphocreatine (PCr) in cerebral grey matter | baseline and 6 months of treatment with Dimethyl Fumarate (DMF)
  PCr levels evaluated by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Changes in ATP in normal appearing white matter (NAWM) | baseline and 6 months of treatment with Dimethyl Fumarate
  ATP levels evaluated by magnetic resonance spectroscopy

OTHER OUTCOMES:
Changes in fatigue | baseline and 6 months of treatment with DMF
  as assessed by Fatigue Severity Scale (FSS), Modified Fatigue Impact Scale (MFIS),
Changes in fatigue | baseline and 6 months of treatment with DMF
  as assessed by Modified Fatigue Impact Scale (MFIS),
Changes in cognition | baseline and 6 months of treatment with DMF
  as assessed by the symbol digit modalities test (SDMT)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spain, MD, MSPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States